CLINICAL TRIAL: NCT04669743
Title: Innate Immunity in Ozone-induced Airway Inflammation in COPD
Acronym: CO3PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-18223
Record Dates: First submitted 2018-12-14; First posted 2020-12-17 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Airway Disease; COPD Exacerbation; Pollution; Exposure; Pollution Related Respiratory Disorder
Keywords: ozone; airway macrophages; air pollution; COPD exacerbation; Phagocytosis; Efferocytosis; Mass cytometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Controlled inhalational challenge to ozone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Population (Experimental): Subjects will be recruited and consented following screening. Subjects will be characterized into cohorts based on presence of COPD and smoking status. All subjects enrolled will be undergoing the same interventions: 1st Bronchoscopy (3 wks pre-exposure), Ozone Exposure, 2nd Bronchoscopy (1 day post-exposure), 3rd Bronchoscopy (5 days post-exposure). Ozone exposure will take place in an exposure chamber.
  Interventions: Other: Ozone exposure

INTERVENTIONS:
Other: Ozone exposure — Exposures will take place at the UCSF Human Exposure Chamber Core Facility. Ozone will be added to the air in the chamber and concentration measured every 30 seconds. Subjects will exercise for two 15-minute intervals of each hour on a cycle ergometer, and will rest for two 15-minute intervals between exercise sessions. The rate of exercise will be individually adjusted to produce a targeted minute ventilation of 15-20 L/min/m2 body surface area. Subjects will be sent home post-exposure and will return to the laboratory on the following day and six days after the exposure for bronchoscopy.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death in the United States. Patients with COPD are routinely exposed to indoor and outdoor air pollution, which appears to cause escalation of their respiratory symptoms, a process called exacerbation, with resulting need to seek medical attention. This research plan proposes to evaluate the impact of lung immune cells in susceptibility to develop exacerbation through an experimental model of inhalational exposure using ambient levels of a component of air pollution (ozone) in COPD patients and longitudinal sampling of their lung immune cells.

DETAILED DESCRIPTION:
A major cause of morbidity and mortality in COPD is exacerbation. The mechanisms underlying COPD exacerbation are poorly understood, but airway innate immune system has been implicated in its development. Air pollution contributes to development of COPD exacerbation, and exposure to ozone, a major component of air pollution, is associated with increased healthcare utilization among patients with COPD. Inhalation of ambient levels of ozone is known to affect airway innate immune system. This proposal sets out to characterize and investigate the role of innate immune system and in particular airway macrophages in ozone-induced COPD exacerbation through establishing an experimental model that employs controlled ozone exposure and longitudinal sampling via bronchoscopy. The research plan proposes to examine human immune cells trafficking in airways during the process of ozone-induced airway injury and inflammation in patients with COPD. The investigator's overall hypothesis is that inhalational challenge to a high ambient level of ozone in patients with COPD provides a safe human model of airway injury with resulting intraluminal shifts in the population and polarization of macrophages to study innate immunity processes relevant to ozone-induced COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

1. No diagnosis of COPD or asthma.
2. No spirometric evidence of airflow obstruction as determined by FEV1/FVC ratio = or >0.7.
3. Less than 1 pack year history of tobacco smoking and no tobacco use within the past 12 months.

Group 2:

1. No diagnosis of COPD or asthma.
2. No spirometric evidence of airflow obstruction as determined by FEV1/FVC ratio = or >0.7.
3. Current smoker with history of at least 20 pack-years smoking.

Group 3:

1. Diagnosis of COPD as determined by GOLD criteria (FEV1/FVC ratio <0.7).
2. COPD severity of GOLD stage II or III (FEV1 >40% predicted).
3. Smoking Status: Former smokers with history of at least 20 pack-years smoking.

Group 4:

1. Diagnosis of COPD as determined by GOLD criteria (FEV1/FVC ratio <0.7).
2. COPD severity of GOLD stage II or III (FEV1 >40% predicted).
3. Smoking Status: Current smokers with history of at least 20 pack-years smoking.

During subject screening visit, Albuterol is used to determine whether the subjects have COPD based on the Global Initiative on Obstructive Lung Diseases (GOLD) criteria. Regardless of whether the subject has reversibility to Albuterol or not, if they have an abnormal ratio after inhalation of Albuterol, they would meet the GOLD criteria for COPD and will be included in the study.

Exclusion Criteria:

1. History of IV drug use or inhalation of recreational drugs other than marijuana:

   A- within the past 20 years. B- more than 100 usage. C- longer than 1 year.
2. COPD severity of GOLD stage IV.
3. Inability to walk briskly or run on treadmill or pedal on ergometer to perform the study-required moderate exercise level (achieve minute ventilation of 15 to 20 L/min/m2 body surface area).
4. Pregnant/breast feeding.
5. Serious and active heart conditions - defined by stable or unstable angina, recent myocardial infarction (within the last 2 years), active congestive heart failure, ischemic cardiomyopathy.
6. Malnourishment - determined by BMI less than 19. If subject has BMI greater or equal to 19, but has a history of malnourishment, study staff will measure albumin level of subject's blood after initial blood draw. Albumin level must be greater than 2.5 mg per deciliter, or subject will be excluded.
7. Liver cirrhosis.
8. History of chronic active Hepatitis B or C
9. On visits where moderate sedation is preformed, subject are required to have an escort home. Inability to secure a ride home will result in the subject being ineligible for the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-04-07 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Changes in prevalence and functional status of alveolar macrophage sub-populations in airway lumen | 4 weeks
  Number of alveolar macrophages (AM) measured by flow cytometry (both absolute numbers and relative percentage of cells)
Changes in prevalence and functional status of monocyte-derived macrophage sub-populations in airway lumen | 4 weeks
  Number of monocyte-derived macrophages (MDM) measured by flow cytometry (both absolute numbers and relative percentage of cells)
Changes in prevalence and functional status of interstitial macrophage sub-populations in airway lumen | 4 weeks
  Number of interstitial macrophages (IM) measured by flow cytometry (both absolute numbers and relative percentage of cells)

SECONDARY OUTCOMES:
Symptomatic responses | 4 weeks
  Evidence for presence of mild exacerbation as measured by changes at or above the level of minimally clinically important difference (MCID) in each of the questionnaire's symptom score, 1-6, for the number of flare-ups in the past 3 years, with 6 being the worst outcome.
Physiologic responses | 4 weeks
  Quantitative changes across ozone exposure in spirometric indices of airflow obstruction
Cardiovascular response using measurement of Heart Rate | 4 weeks
  Cardiovascular outcome of heart rate will be measured for safety assessment before, during, and after ozone exposure. The maximum limit of their heart rate is 80% of their heart rate maximum.
Cardiovascular response using measurement of Blood Pressure | 4 weeks
  Cardiovascular outcome of blood pressure (both systolic and diastolic) will be measured for safety assessment before, during, and after ozone exposure.
Cardiovascular response using measurement of ECG changes | 4 weeks
  Cardiovascular outcomes of electrocardiogram (ECG) changes will be measured for safety assessment before and after ozone exposure. ECG changes, including ST-segment elevation and rhythm abnormalities, will be compared to the baseline ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Arjomandi, M.D., Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No